CLINICAL TRIAL: NCT05712122
Title: Can Stellar Ganglion Blockage be an Alternative Treatment for Refractory Ventricular Arrhythmias?
Brief Title: Stellatar Ganglione Blockage for Ventricular Arrhytmias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cağatay Küçükbingöz, Medical Doctor, Adana City Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 125-85
Record Dates: First submitted 2022-12-17; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- stellat gagnliyon blockadge (Experimental): Ultrasound-guided stellate ganglion blockade and for blockage, the solution was prepared by adding 8 mg dexamethasone, 40 mg lidocaine, and 10 mg bupivacaine to 10 mL with physiological saline.
  Interventions: Procedure: stellate block

INTERVENTIONS:
Procedure: stellate block — stellate blockade effect on Ventricular arrytmia

SUMMARY:
Ventricular tachycardia (VT) and ventricular fibrillation (VF) are life-threatening conditions that increase in frequency over the years. An electrical storm (ES) is defined as the occurrence of 3 or more continuous ventricular arrhythmia. The sympathetic nervous system has an important role in VA and is the target of treatment. Studies show that stellate ganglion blockade (SGB) can reduce cardiac sympathetic tone and is an alternative bridge therapy in VAs. In our study, the investigators preferred to apply a combination of local anesthetic and steroid in the stellate ganglion blocking method to 10 VA patients who were resistant to medical treatment and had an ICD, and we also planned to examine the 6-month follow-up results of the patients.

In our study, USG-guided left stellate ganglion blockade was applied to 10 VA and ES patients with ICD. The 6-month results of the patients were evaluated retrospectively. For blockage, the solution was prepared by adding 8 mg dexamethasone, 40 mg lidocaine, and 10 mg bupivacaine to 10 mL with physiological saline. The success of the procedure was evaluated with the development of Horner's syndrome in the left eye.

DETAILED DESCRIPTION:
In our study, USG-guided left stellate ganglion blockade was applied to 10 VA and ES patients with ICD who were admitted to the Department of Cardiology at Çukurova University between 2020-2021. The 6-month results of the patients were evaluated retrospectively. An electrical storm was defined as 3 episodes of continuous VT/VF or ICD therapy for VT/VF over a 24-hour period. Demographic data and clinical and procedural outcomes of the patients were collected from electronic hospital records. Inpatient telemetry and ICD interrogation logs were reviewed for each patient. Administration of oral and intravenous (IV) anti-arrhythmic drugs (AAD) was recorded for the pre-and post-SGB periods. For our study, approval was taken by the Çukurova University ethics committee on 16.09.2022 with document number 125.

Patient Selection Patients who applied to the Cardiology Department with the diagnosis of VA or ES and did not benefit from antiarrhythmic drug therapy were selected and evaluated by a team of 2 anesthesiologists (cardiothoracic and pain specialists) and 2 cardiologists (1 of whom is an electrophysiology specialist).

All patients received standard treatment modalities based on current American College of Cardiology/American Heart Association/Heart Rhythm Society guidelines for the management of VAs (13). These methods included combinations of therapies for reversible causes (medical treatments, metabolic injuries, myocardial ischemia) beta-blockers, IV AADs, noninvasive programmed stimulation for overrate termination, and ICD programming to optimize anti-tachycardia pacing and minimize shocks. The number of shocks in the last 6 months of the patients selected for the application was checked from the ICD device. Patients with persistent VA storms despite at least 1 antiarrhythmic drug therapy with beta-blocker and catheter ablation for VT were included in the study. After the first injection, VT or VF burden and development of shock were assessed by an implantable cardioverter-defibrillator for 48 hours following the procedure.

Stellat Ganglion Block (SGB) Technique In the operating room, the patients undergoing SGB were hospitalized in the supine position with their heads extended. All patients with intravenous access were monitored with ECG, pulse oximetry, and non-invasive blood pressure in accordance with the guidelines of the American Society of Anesthesiology. Left stellate ganglion blockade was planned for all patients and their heads were turned to the right. The left neck and shoulder of the patient were cleaned with chlorhexidine. The linear (13-6 MHz) USG probe was prepared in accordance with the sterilization conditions. Cervical vertebra level was determined in the neck of the patient with the USG probe at the level of the cricoid cartilage. After visualizing the Chassaignac tubercle, longus coli muscle, carotid, esophagus, and thyroid gland of the C6 vertebra, an 80 mm 22-G, USG compatible (B. Braun Stimuplex Ultra 360) needle was inserted into the medial of the Chassaignac tubercle and towards the front of the prevertebral fascia of the longus Colli muscle using the in-plane technique. After the needle site was confirmed, a negative aspiration test was performed and 10 mL of local anesthetic and steroid mixture was injected (14,15). For blockage, the solution was prepared by adding 8 mg dexamethasone, 40 mg lidocaine, and 10 mg bupivacaine to 10 mL with physiological saline. The success of the procedure was evaluated with the development of Horner's syndrome in the left eye. After the procedure, the patients were taken to the Cardiology Intensive Care Unit and ICD follow-up was performed for 24 hours. The medical treatments of the patients who did not develop a new VA within 24 hours were arranged and they were called for follow-up checkups in the 1st and 6th months. During the check-ups, the number of shocks, the presence of newly developed VA, and whether the patient applied to the emergency department due to VA were followed from the ICD records.

ELIGIBILITY:
Inclusion Criteria:

* Ventricular tachycardia (VT)
* Ventricular fibrillation (VF)
* Electrical storm (ES)

Exclusion Criteria:

* Resistant ventricular arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
ventricular arrhythmia numbers | 6 months
  Determination of 6-month number of new ventricular arrhythmias (In ventricular tachycardia, the heart beats faster, usually 100 or more beats a minute) requirement after stellate ganglion blockade.
ICD shock requirement | 6 months
  Determination of 6-month number of ICD shock (Joule) requirement after stellate ganglion blockade.

CONTACTS AND LOCATIONS:
Locations (1):
- AdanaCityTRH, Adana, Yuregir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meng L, Tseng CH, Shivkumar K, Ajijola O. Efficacy of Stellate Ganglion Blockade in Managing Electrical Storm: A Systematic Review. JACC Clin Electrophysiol. 2017 Sep;3(9):942-949. doi: 10.1016/j.jacep.2017.06.006. PMID 29270467
- [Result] Tian Y, Wittwer ED, Kapa S, McLeod CJ, Xiao P, Noseworthy PA, Mulpuru SK, Deshmukh AJ, Lee HC, Ackerman MJ, Asirvatham SJ, Munger TM, Liu XP, Friedman PA, Cha YM. Effective Use of Percutaneous Stellate Ganglion Blockade in Patients With Electrical Storm. Circ Arrhythm Electrophysiol. 2019 Sep;12(9):e007118. doi: 10.1161/CIRCEP.118.007118. Epub 2019 Sep 13. PMID 31514529
- [Result] Fudim M, Qadri YJ, Waldron NH, Boortz-Marx RL, Ganesh A, Patel CB, Podgoreanu MV, Sun AY, Milano CA, Tong BC, Harpole DH Jr, Mathew JP, Piccini JP. Stellate Ganglion Blockade for the Treatment of Refractory Ventricular Arrhythmias. JACC Clin Electrophysiol. 2020 May;6(5):562-571. doi: 10.1016/j.jacep.2019.12.017. Epub 2020 Feb 26. PMID 32439042

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT05712122/Prot_SAP_000.pdf